CLINICAL TRIAL: NCT01064570
Title: Guidelines for Treatment of Acute Promyelocytic Leukemia
Brief Title: AIDA 2000 Guidelines
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Prof. Franco Mandelli, GIMEMA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIDA2000
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Acute Promyelocytic Leukemia; APL
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: all-trans retinoic acid (ATRA)

SUMMARY:
Prospective use of RT-PCR for PML/RARa might be used to guide a total tehrapy approach in APL, including refined diagnosis, front-line treatment, assessment of response and anticipated salvage therapy for patients who undergo molecular relapse.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 1 years and < 61 years
* Morphologic diagnosis of APL
* PS <= 3
* Presence in leukemic cells at diagnosis of t(15;17), and/or PML/RARa rearrangement by RT-PCR. T
* The presence of additional cytogenetic lesions is not considered an exclusion criterion
* Serum creatinine <=2.5 mg/dL
* Serum bilirubin, alkaline phosphatase, or GOT/ASAT <= 3 times the upper normal limit
* Negative pregnancy test
* Written informed consent

Exclusion Criteria:

* Age >= 61 years
* Prior antileukemic chemotherapy for APL
* Absence of PML-RARa rearrangement after successful RNA extraction and amplification of control gene
* Prior antileikemic chemotherapy for APL
* Presence of a concomitant malignant neoplasm, except basal cell carcinoma Concurrent treatment with cytotoxic chemotherapy or radiotherapy
* Oteher progressive malignant disease. However, secondary acute promyelocytic leukemia following "cured" Hodgkin's disease or otehr cured malignancies may be included, as well as secondary leukemias following other exposure to alkylating agents or radiation for other reasons

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2000-05

PRIMARY OUTCOMES:
Treatment-related toxicity event rate during the ATRA-including consolidation treatment | At the end of the study

SECONDARY OUTCOMES:
Event Free Survival, Molecular and Hematological Disease-Free and Overall Survival in each risk group | At the end of the study
The rates of molecular remission, after consolidation, in each risk group | At the end of the study
Induction morbidity and mortality after the inclusion of the prophylactic measures for the ATRA Syndrome and hemorrhagic complications | At the end of the study
The overall toxicity of induction, consolidation, and maintenance chemotherapy in each risk group | At the end of the study
The impact on survival of a "total" treatment approach for APL including molecular evaluation of minimal residual disease and salvage tehrapy administration at the time of molecular or hematological relapse | At the end of the study

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Unità Operativa Ematologia 1 - Università degli Studi di Bari, Bari
  - Div. di Ematologia IRCCS Policlinico S. Matteo, Pavia
  - A.O Umberto I, Roma

REFERENCES:
- [Background] Breccia M, Mazzarella L, Bagnardi V, Disalvatore D, Loglisci G, Cimino G, Testi AM, Avvisati G, Petti MC, Minotti C, Latagliata R, Foa R, Pelicci PG, Lo-Coco F. Increased BMI correlates with higher risk of disease relapse and differentiation syndrome in patients with acute promyelocytic leukemia treated with the AIDA protocols. Blood. 2012 Jan 5;119(1):49-54. doi: 10.1182/blood-2011-07-369595. Epub 2011 Nov 2. PMID 22049518
- [Result] Lo-Coco F, Avvisati G, Vignetti M, Breccia M, Gallo E, Rambaldi A, Paoloni F, Fioritoni G, Ferrara F, Specchia G, Cimino G, Diverio D, Borlenghi E, Martinelli G, Di Raimondo F, Di Bona E, Fazi P, Peta A, Bosi A, Carella AM, Fabbiano F, Pogliani EM, Petti MC, Amadori S, Mandelli F; Italian GIMEMA Cooperative Group. Front-line treatment of acute promyelocytic leukemia with AIDA induction followed by risk-adapted consolidation for adults younger than 61 years: results of the AIDA-2000 trial of the GIMEMA Group. Blood. 2010 Oct 28;116(17):3171-9. doi: 10.1182/blood-2010-03-276196. Epub 2010 Jul 19. PMID 20644121